CLINICAL TRIAL: NCT03139097
Title: Reference Range Study for the Quantra Analyzer With the Quantra Surgical Cartridge
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-010
Record Dates: First submitted 2017-04-18; First posted 2017-05-03 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Blood samples from healthy volunteers analyzed on the Quantra System.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra Surgical Cartridge

SUMMARY:
This study will establish reference range intervals for the Quantra System, a next-generation diagnostic platform that provides whole blood coagulation testing at the point-of-care.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The Quantra Surgical Cartridge was developed to monitor hemostasis during major surgical procedures in adult patients. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding six parameters that depict the functional status of a patient's coagulation system. In this multi-center, prospective, observational study, blood samples will be obtained from healthy adult volunteers to establish a normal reference range for the test parameters measured by the Quantra System.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years
* Subject is willing to participate and he/she has signed a consent form
* Subject's laboratory coagulation test results at screening are within each test's normal reference range

Exclusion Criteria:

* Subject is younger than 18 years
* Subject has a history of a coagulation disorder
* Subject is pregnant or lactating
* Subject is currently taking medications known to alter coagulation
* Subject had a blood transfusion or surgery within the last month
* Subject has one or more laboratory coagulation test result outside of the normal reference range at screening
* Drug abuse
* Excessive alcohol consumption
* Subject is unable to provide written informed consent
* Subject is incarcerated at the time of the study
* Subject previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult volunteers with normal coagulation function, approximately equal numbers of males and females across three age group categories (18-30, 31-50 and >50 years). The racial and ethnic profiles will be representative of the populations at each site.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Reference range intervals for measurement of Clot Time, Heparinase Clot Time, Clot Stiffness, Fibrinogen Contribution and Platelet Contribution on the Quantra System | Baseline, determined from single blood draw
  Reference range intervals determined in this study from the analysis of blood samples collected from healthy adults will serve as the initial reference ranges for the Quantra test parameters when the Surgical Cartridge is commercially available.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Warren-Ulanch, MD, Principal Investigator — Creedmoor Centre Endocrinology; Charles Greenberg, MD, Principal Investigator — Medical University of South Carolina; Kenichi Tanaka, MD, Principal Investigator — University of Maryland
Locations (3):
- United States (3):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Creedmoor Centre Endocrinology, Raleigh, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No